

## ONDOKUZ MAYIS UNIVERSITY

## KLİNİK ARAŞTIRMALAR ETİK KURULU

Sayı: B.30.2.ODM.0.20.08/120-157-352

16.03.2021

Sayın Prof. Dr. Ramazan AŞÇI

Your biochemistry study+survey study titled "Investigation of the Effects of Lifestyle Changes and Antioxidant Food Supplementation on Semen Antioxidant Capacity, Dna Fragmentation Index and Dna Chromatin Quality in Infertile Patients with Oligoastenoteratozoospermia Detected in Semen Analysis B in the Semen Analysis" that you submitted to our Ethics Committee with the Decision No: OMU KAEK 2021/108 has been examined according to the Clinical Research Ethics Committee Directive in terms of explanations about the reason, approach and method and was decided that there is no ethical objection, that 6-month notifications are made if the duration of the study exceeds 6 months, that the result of the study is notified to us within three (3) months at the latest, unanimously by our Ethics Committee dated 25.02.2021.

I request your information.

Chairman of the Clinical Research Ethics

Committee